CLINICAL TRIAL: NCT00592111
Title: A Comprehensive Study of Clinically Staged Pediatric Hodgkin's Disease: Chemotherapy for All Patients; Supplementary Low Dose Involved Field Irradiation for Selected Patients (CCG 5942)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Children's Cancer Group (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 96-016; CCG 5942; CA42764
Record Dates: First submitted 2007-12-26; First posted 2008-01-11 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-12

CONDITIONS: Pediatric; Hodgkin's Disease
Keywords: Pediatric; Hodgkin's Disease; 96-016
MeSH Terms: conditions — Hodgkin Disease | interventions — CVPPABO protocol; Cyclophosphamide; Vincristine; Procarbazine; Prednisone; Doxorubicin; Bleomycin; Vinblastine; Cytarabine; Etoposide; Granulocyte Colony-Stimulating Factor; Filgrastim

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: COPP/ABV
- 2 (Experimental)
  Interventions: Drug: COPP/ABV
- 3 (Experimental)
  Interventions: Drug: intensive chemo with concurrent growth factor

INTERVENTIONS:
Drug: COPP/ABV — 4 courses of COPP/ABV hybrid
  Other Names: Cyclophosphamide; Vincristine; Procarbazine; Prednisone; Adriamycin; Bleomycin; Vinblastine
  Arms: 1
Drug: COPP/ABV — 6 courses of COPP/ABV hybrid
  Other Names: Cyclophosphamide; Vincristine; Procarbazine; Prednisone; Adriamycin; Bleomycin; Vinblastine
  Arms: 2
Drug: intensive chemo with concurrent growth factor — 6 cycles (2 courses) of intensive chemotherapy with concurrent growth factor
  Other Names: Cyclophosphamide; Vincristine; Procarbazine; Prednisone; Adriamycin; Bleomycin; Vinblastine; Cytosine Arabinoside; Etoposide; G-CSF (Filgrastim)
  Arms: 3

SUMMARY:
Study Hypothesis: Clinical staging without laparotomy/splenectomy is adequate for children and young adults with Hodgkin's disease who receive chemotherapy as a component of treatment.

ELIGIBILITY:
* Age less than 21 years at diagnosis
* Previously untreated, pathologically confirmed diagnosis of Hodgkin's disease.
* Informed patient/parental consent as required by individual institution and in accordance with the Dept of Health and Human Services
* Approval of this protocol by the individual institutional Human Subjects Review Committee.
* Indicate Hodgkin's disease clinical stage.
* Indicate presence or absence of "B" symptoms.
* For Stage I and II disease indicate the following:
* presence or absence of bulk disease
* number of involved nodal regions
* presence or absence of hilar adenopathy

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 1996-03; Primary Completion 1999-02 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Determine the role of adjuvant low dose involved field radiotherapy in pediatric patients with Hodgkin's disease who attain a complete response following initial chemotherapy | Conclusion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Trippett, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Related Info — http://www.mskcc.org